CLINICAL TRIAL: NCT03029871
Title: Phase 1 Trial of Oncolytic Adenovirus-Mediated Cytotoxic Gene Therapy in Combination With Stereotactic Body Radiation Therapy (SBRT) in Clinical Stage 1/11A (T1A-T2B) Non-Small Cell Lung Cancer
Brief Title: Oncolytic Adenovirus-Mediated Gene Therapy for Lung Cancer
Acronym: NSCLC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Benjamin Movsas, M.D. (Other)
Responsible Party: Sponsor-Investigator, Benjamin Movsas, M.D., Chair, Department of Radiation Oncology, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10835
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Non-small Cell Lung Cancer Stage I
Keywords: lung cancer; adenovirus; gene therapy; SBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Intervention Model Description: Nine subjects (3 cohorts, 3 subjects/cohort)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Nine subjects (3 cohorts, 3 subjects/cohort) with medically inoperable stage I/IIA (T1a - T2b) NSCLC with tumors measuring > 2 to ≤ 5 cm will receive a single intratumoral injection of the oncolytic Ad5-yCD/mutTKSR39rep-ADP adenovirus at one of three dose levels (1 x 1011 vp, 3 x 1011 vp, 1 x 1012 vp). Depending on the location of the target lesion, the adenovirus will be injected either transbronchially (central tumors) or percutaneously under computed tomography (CT)-guidance (peripheral tumors). Two days later, subjects will be administered (orally) a 10 day course of 5-fluorocytosine (5-FC) and valganciclovir (vGCV) prodrug therapy along with 48 Gy (4 fractions of 12 Gy) of SBRT. Prior to and following the adenovirus injection, subjects will be administered [18F]-FHBG, a HSV-1 TK substrate, and will undergo PET imaging to quantify HSV-1 TK gene expression.
  Interventions: Biological: Ad5-yCD/mutTKSR39rep-ADP Adenovirus

INTERVENTIONS:
Biological: Ad5-yCD/mutTKSR39rep-ADP Adenovirus — oncolytic adenovirus

SUMMARY:
The primary objective of this phase 1 trial is to determine the dose-dependent toxicity and maximum tolerated dose (MTD) of oncolytic adenovirus-mediated cytotoxic gene therapy in combination with SBRT in medically inoperable stage I/IIA (T1A - T2B) NSCLC. To accomplish this objective, 9 subjects will be enrolled in the study. We hypothesize that the combined treatment will demonstrate acceptable toxicity, and that it will be feasible to quantify adenovirus-mediated HSV-1 TK gene expression in the lung by PET. This phase 1 trial will lay the foundation for a follow-up phase 2 trial designed to examine efficacy.

DETAILED DESCRIPTION:
Nine subjects (3 cohorts, 3 subjects/cohort) with medically inoperable stage I/IIA (T1a - T2b) NSCLC with tumors measuring > 2 to ≤ 5 cm will receive a single intratumoral injection of the oncolytic Ad5-yCD/mutTKSR39rep-ADP adenovirus at one of three dose levels (1 x 1011 vp, 3 x 1011 vp, 1 x 1012 vp). Depending on the location of the target lesion, the adenovirus will be injected either transbronchially (central tumors) or percutaneously under computed tomography (CT)-guidance (peripheral tumors). Two days later, subjects will be administered (orally) a 10 day course of 5-fluorocytosine (5-FC) and valganciclovir (vGCV) prodrug therapy along with 48 Gy (4 fractions of 12 Gy) of SBRT. Prior to and following the adenovirus injection, subjects will be administered [18F]-FHBG, a HSV-1 TK substrate, and will undergo PET imaging to quantify HSV-1 TK gene expression. Toxicity assessments will occur twice a week for the first 2 weeks and then at scheduled follow-up visits through 60 months. The primary endpoint is toxicity. Secondary endpoints include 1) tumor (radiological) response, 2) local, regional, and distal tumor control, 3) progression-free and overall survival, and 4) quality of life. Exploratory endpoints include 1) intensity, persistence, and biodistribution of HSV-1 TK gene expression, and 2) association of select serum biomarkers with toxicity and tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of NSCLC.
* Clinical stage I/IIA (T1a - T2b; AJCC Staging 7th edition) with a tumor size > 1 cm to ≤ 6 cm in diameter (long axis) based on the following minimum diagnostic workup:

Note: Subjects may have M0 or MX status (e.g., lung nodules that are being observed). Known M1 disease is excluded. Subjects may have only one target lesion for SBRT.

* Evaluation at lung multi-disciplinary tumor board with recommendation for SBRT within 12 weeks of registration.
* Whole body positron emission tomography (PET/CT) scan within 12 weeks of registration using [18F]-FDG with adequate visualization of the primary tumor and draining lymph node basins in the hilar and mediastinal regions.

Mediastinal lymph node sampling by any technique is allowed but not required. Subjects with > 1.5 cm mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsies of abnormally identified areas are negative for cancer.

* Zubrod Performance Status 0 - 2 with 4 weeks of registration.
* Age ≥ 18.
* Subjects must have adequate baseline organ function, as assessed by the following laboratory values, within 30 days before initiating the study therapy:
* Adequate renal function with serum creatinine ≤ 1.5 mg/dL or creatinine clearance >50 mL/min/m2.
* Platelet count > 100,000/μL.
* Absolute neutrophil count > 1,000/μL.
* Hemoglobin > 10.0 g/dL.
* Bilirubin > 1.5 mg/dL
* AST/SGOT and ALT/SGPT < 3.0 times upper limit of normal (ULN).
* Negative serum or urine pregnancy test within 72 hours prior to the adenovirus injection for women of childbearing potential.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout and for 60 days beyond the treatment phase of the study.
* Subjects must possess the ability to give informed consent and express a willingness to meet all of the expected requirements of the protocol for the duration of the study.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (e.g., carcinomas in situ of the breast, oral cavity, or cervix are permissible). Subjects with previous lung cancer are permitted if the subject is disease-free for a minimum of 2 years or if this is a solitary recurrence in the lung measuring > 2 cm and ≤ 5 cm after surgery.
* Any known metastatic disease. Subjects may have MX status (e.g., lung nodules that are being observed).
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Prior chemotherapy for the study cancer.
* Plans for the subject to receive other local therapy (including standard fractionated radiotherapy and/or surgery and/or other local ablative therapies) while on this study, except in the case of disease progression.
* Plans for the subject to receive systemic therapy (including standard chemotherapy or biologic targeted agents), while on this study, except in the case of disease progression.
* Acute infection. Acute infection is defined by any viral, bacterial, or fungal infection that requires specific therapy within 72 hours of initiation of the study therapy.
* Previous history of liver disease including hepatitis.
* Immunosuppressive therapy including systemic corticosteroids. Use of inhaled and topical corticosteroids is permitted.
* Impaired immunity or susceptibility to serious viral infections.
* Allergy to any product used in the protocol.
* Serious medical or psychiatric illness or concomitant medication, which, in the judgment of the principal investigator, might interfere with the subject's ability to respond to or tolerate the treatment or complete the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity and maximum tolerated dose | 60 days
  Treatment-related adverse events (CTCAE v4.03)

SECONDARY OUTCOMES:
Tumor response | 3 months to 5 years
  RECIST
Survival | 3 months to 5 years
  Progression-free and overall
Quality of Life | 3 months to 5 years
  FACT-TOI (Functional Assessment of Cancer Therapy-Trial Outcome Index)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No